CLINICAL TRIAL: NCT05788744
Title: Implementing Non-invasive Circulating Tumor DNA and Circular DNA Analysis in Patients With Localized Pancreatic Cancer to Optimize the Pre- and Postoperative Treatment: Predicting Recurrence and Survival and Changing Prognosis Over Time
Brief Title: Implementing ctDNA and Circular DNA in Patients With Localized Pancreatic Cancer
Acronym: CIRCPAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Collaborators: Aarhus University Hospital (Other); University of Copenhagen (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Prof. Julia Sidenius Johansen, Professor, Copenhagen University Hospital at Herlev
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CIRCPAC
Record Dates: First submitted 2022-11-23; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Resectable Pancreatic Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Experimental (Experimental): Patients will receive surveillance with liver enzymes, CA 19-9, history, clinical evaluation of signs of recurrence (e.g. weight loss, abdominal pain or fatigue) in combination with analysis of plasma ctDNA (90 ml blood drawn per visit) every 3 months until disease progression or up to 36 months. If plasma ctDNA is positive the patient will have a CT scan (thorax and abdomen) and EUS every 3 months for 2 years and then every 6 months until disease recurrence or up to 36 months. If plasma ctDNA is negative the patient will have CT scan of thorax and abdomen and EUS every 6 months until disease recurrence or up to 36 months. Plasma eccDNA will be determined at the same time as ctDNA but a positive eccDNA result will not be informed to the patients.
  Interventions: Diagnostic Test: ctDNA
- B: Control (No Intervention): Patients will receive surveillance until recurrence according to current Danish guidelines with liver enzymes, history and clinical evaluation every 3 months for two years and then every 6 months until 36 months. If an increase in liver enzymes is seen or clinical signs of recurrence (e.g. weight loss, abdominal pain or fatigue) patients will have a CT scan of thorax and abdomen. Blood samples (90 ml blood per visit) will be collected at the same time points as blood is drawn for liver enzymes (i.e. every 6 months until 36 months) for later analysis at the end of study of plasma ctDNA and eccDNA. These measurements will serve to enable post-trial comparison of oncological outcomes for the two arms.

INTERVENTIONS:
Diagnostic Test: ctDNA — ctDNA guided surveillance
  Other Names: eccDNA
  Arms: A: Experimental

SUMMARY:
The goal of this clinical trial is to investigate if plasma ctDNA and eccDNA before resection for suspicion of pancreatic ductal adenocarcinoma (PDAC) can predict early recurrence and overall survival, and to investigate if plasma ctDNA combined with CT scan and endoscopic ultrasound surveillance increases the median overall survival compared with standard-of-care surveillance.

DETAILED DESCRIPTION:
The aim of the CIRCPAC study is to evaluate if plasma ctDNA from patients scheduled for surgical resection of PDAC can identify patients who will benefit from surgery and if plasma ctDNA can identify recurrence earlier and improve the survival and quality of life of the patients compared with standard-of-care surveillance.

Patients operated for PDAC will be included in this Danish multicenter study including an observational study (Sub-study 1: 700 patients) and an interventional randomized trial (Sub-study 2: 410 patients).

In Sub-study 1, patients will have blood samples drawn prior to surgery, 4 weeks after surgery, and 6 months after surgery.

In Sub-study 2, patients without recurrence 4 months after surgery, will be randomized in a 1:1 manor to an experimental arm (arm A) with ctDNA guided surveillance, or to a control arm (B) with standard surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Sub-study 1: Suspicion of PDAC tumor stage I-III, scheduled for pancreatic resection, with or without preoperative neoadjuvant chemotherapy.
* Sub-study 2: .

  * PDAC tumor stage I-III
  * Has received intended curative resection (R0/R1) of PDAC
  * No signs of local recurrence or metastatic disease at a CT scan 4 months after the operation

Exclusion Criteria:

* Other cancers (excluding skin cancer other than melanoma) later than 3 years before inclusion
* Patients who are unlikely to comply with the protocol, inability to return for subsequent visits) and/or otherwise considered by the Investigator to be unlikely to complete the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Sub-study 1 ctDNA | 36 months
  Preoperative plasma ctDNA levels before PDAC resection predicting early recurrence.
Sub-study 1 eccDNA | 36 months
  Preoperative plasma eccDNA levels before PDAC resection predicting early recurrence.
Sub-study 2 ctDNA DFS | 3 years from surgery for PDAC
  Number of patients with recurrence assessed by ctDNA
Sub-study 2 ctDNA OS | 3 years from surgery for PDAC
  Overall survival of patients in arm A compared with patients in Arm B
Sub-study 2 eccDNA | 3 years from surgery for PDAC
  Number of patients with recurrence assessed by eccDNA

CONTACTS AND LOCATIONS:
Overall Officials: Julia S Johansen, MD, Principal Investigator — Copenhagen University Hospital - Herlev and Gentofte
Locations (5):
- Denmark (5):
  - Aalborg Universitetshospital, Aalborg
  - Aarhus Universitetshospital, Aarhus
  - Copenhagen University Hospital - Rigshospitalet, Copenhagen
  - Copenhagen University Hospital - Herlev and Gentofte, Herlev
  - Odense Universitetshospital, Odense

IPD SHARING:
Plan to Share IPD: No
If sharing through anonymization is possible, then yes.